CLINICAL TRIAL: NCT02737423
Title: Vitamin D for the Treatment of Painful Diabetic Neuropathy
Brief Title: Vitamin D Treatment for Painful Diabetic Neuropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baqai Institute of Diabetology and Endocrinology (Other)
Responsible Party: Principal Investigator, Abdul Basit, Professor of Medicine, Director of Baqai Institute of Diabetology and Endocrinology, Baqai Institute of Diabetology and Endocrinology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: BIDE-12/2014
Record Dates: First submitted 2016-02-01; First posted 2016-04-14 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-04

CONDITIONS: Diabetic Neuropathy
MeSH Terms: conditions — Diabetic Neuropathies | interventions — Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- vitamin D (Experimental): single IM dose 600,000 IU of cholecalciferol
  Interventions: Drug: cholecalciferol

INTERVENTIONS:
Drug: cholecalciferol — Effect of Vitamin D on the symptoms of diabetic neuropathy
  Other Names: Vitamin D3

SUMMARY:
The main objective of the study is to assess the effect of vitamin D treatment on painful diabetic neuropathy in Pakistan.

This is a prospective study of diabetic patients with a DN score ≥ 4, administered a single dose of 600,000 IU of Vitamin D.

All diabetic patients (type 1 and type 2) at the screening visit were considered eligible to participate in the study. The change in painful diabetic neuropathy scores was assessed using DN4 Neuropathic Pain Diagnostic Questionnaire and SF - MPQ for all participants at each visit.

DETAILED DESCRIPTION:
Background Painful diabetic neuropathy (DPN) is common in patients with long-standing diabetes mellitus. The prevalence of neuropathy approaches 50% in those with diabetes for 25 years. Among patients with neuropathy, 11.6% with type 1 diabetes and 32.1% with type 2 diabetes have neuropathic pain. In our recent observational study of a large cohort of diabetic patients from primary care in northwest England (n = 15,692), painful diabetic neuropathy (PDN), assessed using the neuropathy symptom score (NSS) and neuropathy disability score (NDS) (NSS >/=5 and NDS >/=3) was 21%, and the prevalence of painful symptoms (NSS >/=5) was 34%. Despite less neuropathy in South Asians (14%) compared to Europeans (22%) (P < 0.0001), painful symptoms were greater in South Asians (38 vs. 32%, P < 0.0001) and they maintained a 50% increased risk of painful neuropathy symptoms (P < 0.0001).

The potential for an association between vitamin D and a beneficial effect on neuropathy is based on experimental data which has shown that vitamin D3 can upregulate NGF and the products of its neuronal target genes resulting in an improvement in experimental diabetic neuropathy. Vitamin D insufficiency has recently been associated with retinopathy and self-reported peripheral neuropathy symptoms even after adjusting for demographic factors, obesity, comorbidities, use of medications for neuropathy and diabetes duration and glycemic control. Of course, there may be some overlap between the symptoms associated with vitamin D deficiency and diabetic neuropathy, which may partly explain the excess painful symptoms we have observed in Asians, particularly as the latter have excess vitamin D deficiency.

The preliminary data suggests there is an urgent need to undertake a blinded placebo-controlled randomised trial of vitamin D3 in the treatment of diabetic peripheral neuropathy.

Aims:

* To see the association of Serum Vitamin D3 levels in type 2 diabetic subjects with Painful neuropathy
* Effect of intervention through injectable Vitamin D3 on Painful diabetic neuropathy Study Design The study is a single centre, single (patient)-blinded, evaluation of injectable cholecalciferol in the treatment of painful diabetic neuropathy.

Study Drug: Injectable cholecalciferol (inj. Vitamin D3 600,000 IU).

1. Sample size = 165 type 2 diabetic subjects
2. Recruitment time = 12 weeks
3. Treatment duration = 12 weeks

Data Analysis and Statistical Considerations:

The normality of the data will be assessed and if the data are severely non-normal, log transformations will be considered. The primary analysis will compare the change from baseline without an alpha adjustment for the multiple comparisons. Comparisons within each treatment group across time will also be considered. The analysis will be performed with Last Observation Carried Forward (LOCF).

Assessment during the Treatment Period:

* Change from baseline in DN4
* Change from baseline in SF-MPQ
* Change from baseline in NeuroQol
* Change from baseline in serum 25 (OH) D, serum corrected calcium; parathyroid hormone, serum phosphate; serum ALP
* Change from baseline in HbA1c; fasting glucose; CBC, urea, creatinine, electrolytes, urine DR, fasting lipid profile

ELIGIBILITY:
Inclusion Criteria:

* All patients with type 1 or type 2 diabetes aged 18 to 80 years
* Patient has a diagnosis of painful diabetic neuropathy and reports symmetrical painful symptoms in distal extremities for a period of 1-5 years prior to the study, and symptoms were attributable to DPN
* HbA1c level ≤ 11% at the screening visit were considered eligible to participate in the study.

Exclusion Criteria:

* Patients with renal impairment or hypo or hyperthyroidism,
* Patients currently taking vitamin D supplementation or anti - epileptic or anti - tuberculosis medication,
* Patients with a previous or current history of primary or tertiary hyperparathyroidism, hypercalcemia, psychiatric disorder, alcohol dependency, Hepatitis B or C, HIV infection and peripheral neuropathy due to a non-diabetic cause
* Pregnant or breast feeding female patients
* Patients allergic to nuts or any nut products and patients participating in any other interventional research trial were excluded from the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2012-06; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Improvement in painful diabetic neuropathy by the use of vitamin D Injections (600,000 IU) assessed with the DN4 Neuropathic Pain Diagnostic Questionnaire | 5 months
  DN4 Neuropathic Pain Diagnostic Questionnaire contains six questions which reflect positive symptoms for pain i.e. question 1, 2, 3, 4, 5 and 10 (sensations of burning, painful cold, electric shocks, tingling, pins & needles and brushing).

SECONDARY OUTCOMES:
Improvement in painful diabetic neuropathy by the use of vitamin D Injections (600,000 IU) assessed with the SF-Mac Gill Pain Questionnaire. | 5 months
  SF-Mac Gill pain questionnaire was evaluated to establish the sensory dimensions of pain which included pain sensations like throbbing, shooting, stabbing, sharp, cramping, gnawing, hot burning, aching, heavy, tender and splitting and effective dimensions of the pain experience which included sensations like tiring-exhausting, sickening, fearful and punishing-cruel.

CONTACTS AND LOCATIONS:
Overall Officials: Abdul Basit, MRCP, Principal Investigator — Baqai Institute of Diabetology and Endocrinology, Baqai Medical University

IPD SHARING:
Plan to Share IPD: Undecided